CLINICAL TRIAL: NCT02267070
Title: Enhancing Cognitive Training Through Exercise After a First Schizophrenia Episode
Acronym: CT&E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH102529-01 (NIH); R34MH102529 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2014-10-17 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: cognitive training; aerobic exercise; neurotrophic factors; randomized controlled trial
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Case Management; Cognitive Training; Cognitive Remediation; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training and Exercise (Experimental): 24 weeks of systematic computerized cognitive training, 4 hours per week, plus aerobic exercise, four 30 minute sessions per week. The first 12 weeks involves neurocognitive training, using auditory training exercises from Posit Science Brain HQ. The 2nd 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. Aerobic exercise occurs as two 30-minute sessions at the clinic and two at home weekly. Intensity of aerobic exercise is tailored to maintain an individualized target heart rate zone and is monitored by a heart rate recorder. A weekly one-hour Bridging Skills Group is designed to aid generalization of training to everyday life situations. All members receive individual case management and supportive psychotherapy, and family psychoeducation.
  Interventions: Behavioral: Case management and supportive psychotherapy; Behavioral: Family psychoeducation; Behavioral: Cognitive training; Behavioral: Aerobic exercise
- Cognitive Training (Active Comparator): 24 weeks of systematic computerized cognitive training, 4 hours per week, plus aerobic exercise, four 30 minute sessions per week. The first 12 weeks involves neurocognitive training, using auditory training exercises from Posit Science Brain HQ. The 2nd 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. A weekly one-hour Bridging Skills Group is designed to aid generalization of training to everyday life situations. All members receive individual case management and supportive psychotherapy, and family psychoeducation.
  Interventions: Behavioral: Case management and supportive psychotherapy; Behavioral: Family psychoeducation; Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Case management and supportive psychotherapy — An individual therapist will provide weekly case management and therapy targeting the individual psychological problems and everyday functioning needs of the patient
Behavioral: Family psychoeducation — All immediate family members will be invited to family psychoeducation sessions.
Behavioral: Cognitive training — The Cognitive Training and Exercise intervention involves 24 weeks of systematic computerized cognitive training, 4 hours per week, plus aerobic exercise, four 30 minute sessions per week. The first 12 weeks involves neurocognitive training, using auditory training exercises from Posit Science Brain HQ. The second 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. A weekly one-hour Bridging Skills Group with other members of the treatment condition is designed to aid generalization of training to everyday life situations.
  Other Names: cognitive remediation
Behavioral: Aerobic exercise — Aerobic exercise occurs as two 30-minute sessions at the clinic and two at home weekly. Intensity of aerobic exercise is tailored to maintain an individualized target heart rate zone and is monitored by a heart rate recorder.
  Other Names: physical exercise
  Arms: Cognitive Training and Exercise

SUMMARY:
This is a randomized controlled 6-month trial of the efficacy of a novel intervention combining neuroplasticity-based cognitive training with aerobic exercise, compared to the same systematic cognitive training alone. The primary treatment targets are overall cognitive deficit level and independent living skills. The investigators hypothesize that combining neuroplasticity-based computerized cognitive training and neurotrophin-enhancing physical exercise will produce large cognitive and functional improvements, even relative to cognitive training alone. Adding aerobic exercise to a cognitive training program will have the additional benefit of helping to ameliorate medication side effects, reduce the risk for developing metabolic syndrome, and help to prevent the deterioration in physical health that usually follows the onset of schizophrenia and its pharmacologic treatment. The investigators target the period shortly after a first episode of schizophrenia to maximize the generalization of cognitive improvement to functional outcome, before chronic disability is established.

DETAILED DESCRIPTION:
The Cognitive Training and Exercise intervention involves 24 weeks of systematic computerized cognitive training, 4 hours per week, plus aerobic exercise, four 30 minute sessions per week. The first 12 weeks involves neurocognitive training, using auditory training exercises from Posit Science Brain HQ. The second 12 weeks involves social cognitive training, using the Posit Science SocialVille modules. Aerobic exercise occurs as two 30-minute sessions at the clinic and two at home weekly. Intensity of aerobic exercise is tailored to maintain an individualized target heart rate zone and is monitored by a heart rate recorder. A weekly one-hour Bridging Skills Group with other members of the treatment condition is designed to aid generalization of training to everyday life situations.

ELIGIBILITY:
Inclusion Criteria:

1. a first episode of a psychotic illness that began within the past two years;
2. a diagnosis by Diagnostic and Statistical Manual of Mental Disorders of schizophrenia, schizoaffective disorder, mainly depressed type, or schizophreniform disorder;
3. between 18 and 45 years of age;
4. sufficient acculturation and fluency in the English language to avoid invalidating research measures of thought, language, and speech disorder or of verbal cognitive abilities; and
5. residence within commuting distance of the Aftercare Research Program at the University of California, Los Angeles.

Exclusion Criteria:

1. evidence of a known neurological disorder (e.g., epilepsy) or significant head injury;
2. evidence of alcohol or substance use disorder within the six months prior to the first episode and evidence that substance abuse triggered the psychotic episode or makes the schizophrenia diagnosis ambiguous;
3. mental retardation, i.e. premorbid intelligence quotient less than 70.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) overall composite score | 6 months
  The overall composite score from the MCCB is a summary of cognitive performance across seven domains.

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor (BDNF) | 6 months
  BDNF is a principal growth factor known to mediate the effects of exercise in the brain.
Cardiorespiratory fitness | 6 months
  Cardiorespiratory fitness, a secondary physical health outcome variable, will be measured using a ramped version of the traditional Bruce treadmill protocol.
University of California, San Diego (UCSD) Performance-Based Skills Assessment (UPSA) | 6 months
  The UCSD Performance-Based Skills Assessment (UPSA)assesses five all-purpose skills that are important for functioning in the community: general organization, finance, social/communications, transportation, and household chores.
Facial Emotion Identification Test | 6 months
  The Facial Emotion Identification Test involves choice of emotions in facial expressions of 6 different emotions (happy, sad, angry, afraid, surprised, disgusted) plus neutral expressions.
Prosody Task | 6 months
  The Prosody Task involves identifying emotions in audio recordings of male and female actors portraying 5 emotions.
Global Functioning Scale | 6 months
  A 10-point rating scale to evaluate role and social functioning
Modified Social Adjustment Scale - Work Outcome | 6 months
  A measure of the quantity and type of work at a job, school, or in the home
Independent Living Skills Survey | 6 months
  The Independent Living Skills Survey is a 76-item measure based on patient interview, which provides a more detailed assessment of 11 daily living skill domains
Quality of Life Scale | 6 months
  The Quality of Life scale135, a 53-item interview-based inventory, assesses a patient's subjective satisfaction in several key domains
Role Functioning Scale: Work Productivity, Social Relationships, Family Relationships | 6 months
  The Role Functioning Scale is a global clinician-rated measure of everyday functioning in several domains.
Independent Living rating from Role Functioning Scale | 6 months
  The Independent Living rating assesses daily living skills and extent of living independently based on a clinician interview.

CONTACTS AND LOCATIONS:
Overall Officials: Keith H Nuechterlein, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Le TP, Ventura J, Ruiz-Yu B, McEwen SC, Subotnik KL, Nuechterlein KH. Treatment engagement in first-episode schizophrenia: Associations between intrinsic motivation and attendance during cognitive training and an aerobic exercise program. Schizophr Res. 2023 Jan;251:59-65. doi: 10.1016/j.schres.2022.12.018. Epub 2022 Dec 26. PMID 36577235
- [Derived] McEwen SC, Jarrahi B, Ventura J, Subotnik KL, Nguyen J, Woo SM, Nuechterlein KH. A combined exercise and cognitive training intervention induces fronto-cingulate cortical plasticity in first-episode psychosis patients. Schizophr Res. 2023 Jan;251:12-21. doi: 10.1016/j.schres.2022.12.001. Epub 2022 Dec 15. PMID 36527955
- [Derived] Nuechterlein KH, McEwen SC, Ventura J, Subotnik KL, Turner LR, Boucher M, Casaus LR, Distler MG, Hayata JN. Aerobic exercise enhances cognitive training effects in first-episode schizophrenia: randomized clinical trial demonstrates cognitive and functional gains. Psychol Med. 2023 Jul;53(10):4751-4761. doi: 10.1017/S0033291722001696. Epub 2022 Aug 8. PMID 36047035